CLINICAL TRIAL: NCT01603758
Title: Reverse Cholesterol Transport in Humans
Brief Title: Physiological Study of Human Cholesterol Metabolism and Excretion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Richard E. Ostlund Jr., MD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Richard E. Ostlund Jr., MD, Professor of Medicine, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 201110042; R01HL108160 (NIH)
Record Dates: First submitted 2012-05-18; First posted 2012-05-23 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Heart Disease; Cardiovascular Disease; Dyslipidemia; Disorder of Cholesterol Metabolism
Keywords: Cholesterol; Spectrometry, mass; Deuterium; Kinetics; Cholesterol absorption; Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Dyslipidemias; Arachnodactyly | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observational Arm (No Intervention): Cholesterol metabolic parameters will be measured in 100 subjects in an observational study. Results will be related to circulating biomarkers and carotid intima-media thickness.
- Ezetimibe Interventional Arm (Placebo Comparator): Cholesterol metabolic parameters will be measured before and after ezetimibe or placebo intervention. Changes due to ezetimibe will be determined
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe 10 mg/day or placebo will be given for 6 weeks
  Other Names: Zetia
  Arms: Ezetimibe Interventional Arm

SUMMARY:
The underlying hypothesis is that whole body cholesterol - including cholesterol present in tissues that cannot be measured by standard blood tests - is related to heart disease risk. Endogenous cholesterol will be labeled with an intravenous infusion of one type of cholesterol tracer and dietary cholesterol will be labeled with another. These tracers will be used to measure how fast cholesterol is synthesized and excreted using mass spectrometry to distinguish the tracers. Data will be related to circulating biomarkers (blood tests) and to the thickness of the lining of the carotid artery. The effect of the drug ezetimibe on these processes will also be determined. Successful completion of this study will give us more knowledge about cholesterol metabolism that may be useful in designing new drugs and treatments for patients with heart disease, especially those that are already receiving maximum amounts of current medications.

DETAILED DESCRIPTION:
The central hypothesis of this proposal is that reverse cholesterol transport is related to coronary heart disease (CHD) risk. It is complementary to the concept that reduction of cholesterol biosynthesis with statin drugs prevents CHD, but it focuses on whole body cholesterol metabolism and kinetic cholesterol transport rather than on static levels of circulating lipoproteins. Although this is an old idea, it has not been adequately tested in humans because of lack of suitable methods. In this proposal we will apply innovative stable isotope and mass spectroscopic technology to study reverse cholesterol transport in human subjects. The first specific aim is to improve the preparation of intravenous deuterated cholesterol tracer, a critical limiting element in the study of whole body cholesterol metabolism. The second aim is to use that intravenous tracer, along with a different oral tracer, to partition fecal cholesterol into excreted endogenous cholesterol, unabsorbed dietary cholesterol and newly-synthesized cholesterol derived from the liver and intestine. Measurements will be made during consumption of a controlled diet provided by the metabolic kitchen. The pool size of the rapidly-mixing body cholesterol pool will be measured along with the fractional rate of cholesterol catabolism. These direct measures of reverse cholesterol transport will be correlated with plasma biomarkers and with metabolic covariates. The relation of reverse cholesterol transport to carotid intima-media thickness will be determined. The third specific aim will use similar methods to study the mechanism of action for the widely-used drug ezetimibe. The fractional rate of endogenous cholesterol excretion and the rate of plasma cholesterol turnover will be determined in two periods, one with drug and one with placebo treatment. This work represents a new direction for cholesterol research with the potential to develop new and complementary methods of reducing CHD risk that can be added to diet and statin drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aim II. 100 subjects aged 30-80 with stable medical and/or surgical illnesses.
* Aim III. 30 subjects age 18-80 with LDL cholesterol <190, fasting triglycerides<250 and stable medical or surgical illnesses.

Exclusion Criteria:

* Aim II. Subjects taking ezetimibe, bile acid sequestrants or with gastrointestinal or liver disease will be excluded since these may affect whole body cholesterol metabolism.
* Subjects with coronary heart disease or other medical illnesses will not be excluded if medically stable.
* Adults under age 30 and children will be excluded because in our current database there is no relation between carotid intima-media thickness and cardiovascular risk factors in this younger group.
* Aim III. Individuals have risk factors for coronary heart disease that mandate drug treatment according to the National Cholesterol Education Program guidelines will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Fractional Excretion of Endogenous Cholesterol | 4 years
  The fractional rate of endogenous cholesterol excretion will be measured and related to circulating biomarkers and carotid intima-media thickness (Aim #2) or the change in fractional endogenous cholesterol excretion after treatment with ezetimibe will be determined (Aim #3)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Ostlund, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared subject to IRB and HIPAA restrictions.

REFERENCES:
- [Derived] Lin X, Racette SB, Ma L, Wallendorf M, Davila-Roman VG, Ostlund RE Jr. Endogenous Cholesterol Excretion Is Negatively Associated With Carotid Intima-Media Thickness in Humans. Arterioscler Thromb Vasc Biol. 2017 Dec;37(12):2364-2369. doi: 10.1161/ATVBAHA.117.310081. Epub 2017 Oct 5. PMID 28982667
- [Derived] Lin X, Racette SB, Ma L, Wallendorf M, Ostlund RE Jr. Ezetimibe Increases Endogenous Cholesterol Excretion in Humans. Arterioscler Thromb Vasc Biol. 2017 May;37(5):990-996. doi: 10.1161/ATVBAHA.117.309119. Epub 2017 Mar 9. PMID 28279967